CLINICAL TRIAL: NCT06690125
Title: Attention, Awareness, and Multisensory Integration in Patients with Unilateral Spatial Neglect Following Stroke
Brief Title: Multisensory Integration and Cognitive Awareness in Post-Stroke Unilateral Spatial Neglect
Status: Completed | Type: Observational
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Valentina Varalta, Doctor, Universita di Verona
Other Study IDs: 1975CESC
Record Dates: First submitted 2024-10-30; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2018-11

CONDITIONS: Neglect, Hemispatial; Stroke Acute
Keywords: neglect; attention; awareness; multisensory integration
MeSH Terms: conditions — Perceptual Disorders; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with right hemisphere stroke (Without USN)
  Interventions: Diagnostic Test: Classical and computerized assessment
- Patients with right hemisphere stroke (With USN)
  Interventions: Diagnostic Test: Classical and computerized assessment

INTERVENTIONS:
Diagnostic Test: Classical and computerized assessment — Patients with right hemisphere stroke will undergo a battery of standardized paper-based tests, as part of routine clinical practice, including cognitive assessments.
  Additionally, they will complete computerized tests involving the presentation of unisensory (Auditory or Visual Stimuli) and multisensory stimuli (visual and auditory stimuli)

SUMMARY:
The primary aim of this study is to investigate whether multisensory integration (MSI) mechanisms observed in patients with right hemisphere lesions without neglect remain intact compared to patients with Unilateral Spatial Neglect (USN).

This study also allows for a direct comparison between results from paper-based tests and computerized tests, as well as between patients with right hemisphere lesions without neglect and USN patients. The secondary objectives are:

To compare these results in order to obtain a more refined definition of USN at both the unisensory level (as computerized tests are rarely used in hospital settings but have proven effective in diagnosing USN) and the multisensory level (since USN is not generally tested in the auditory modality).

To measure eye movements in all patients in the study, as this can provide useful information for characterizing patient deficits.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in the study if they have:
* Right hemisphere stroke
* Presence of USN assessed through the Apple Cancellation
* Age between 18 and 85 years
* Signed informed consent
* Both male and female participants

As a control group, patients will also be included if they have:

* Right hemisphere stroke
* Absence of USN assessed through the Apple Cancellation
* Age between 18 and 85 years
* Signed informed consent
* Both male and female participants.

Exclusion Criteria:

* Both patients with USN and control patients will be excluded if they:
* Are minors
* Are unable to give their consent to participate in the study
* Have significant language deficits (production and comprehension) (e.g., unable to give a verbal response or understand instructions)
* Have hemianopia
* Have severe hearing impairments that cannot be corrected (e.g., with hearing aids)
* Have severe uncorrected visual impairments (e.g., glaucoma)
* Have a history of psychiatric disorders or substance abuse.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke who have right hemisphere lesions and showed USN.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Multisensory Computerized Test | The assessment is conducted within a week of admission to the ward.
  The test is structured into three tasks that characterize the patient's deficits through visual and auditory stimuli.
  In Task 1, 100 light items are presented in two blocks of 50, while in Task 2, the patient interacts with 36 sound items in a single block. During these tasks, the patient, seated in front of the computer, must localize the sources of light and sound. The lights are generated on the screen using software like MATLAB, while sounds come from speakers mounted on the screen. The patient's responses are recorded via a microphone and noted by the experimenter using the keyboard.
Multisensory Computerized Test | Is conducted over a total of three different days, during which the patient will complete Task 3 in three separate sessions, one for each day.
  In Task 3, the presentation occurs simultaneously, with 360 items distributed across 12 blocks of 30 items each, repeated over three days. In this case as well, the patient must localize the sources of light and sound. This integrated approach allows for a thorough evaluation of sensory localization abilities and analyzes the interaction between visual and auditory stimuli in the patient.

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE) | The assessment is conducted within a week of admission to the ward.
  (Range: 0-30; higher score=best performance).
Apple Cancellation Test | The assessment is conducted within a week of admission to the ward.
  The Apple Cancellation Test is a neuropsychological assessment that evaluates visual attention and neglect, both egocentric and allocentric, particularly in patients with brain injuries. During the test, participants are presented with a sheet containing a grid with 15 apples per cell: three large (one without an opening, one with an opening on the left, and one with an opening on the right) and 12 small apples (four without openings, four with openings on the left, and four with openings on the right). Participants must cancel the target apples within a set time frame.
  The total score is based on the number of targets canceled, with a maximum of 50 apples. Additionally, an asymmetry score for egocentric neglect is calculated, representing the difference between the number of targets selected on the right side (boxes 1-4) and the number of targets selected on the left side (boxes 7-10). Higher scores indicate better performance, while lower scores may suggest difficulties in attentio
Line Bisection Test | The assessment is conducted within a week of admission to the ward.
  In the Line Bisection Test, the patient is asked to mark the midpoint on a series of lines. For each line, a score is assigned that ranges from 0 to 3: a score of 0 indicates an inaccurate indication, while higher scores (up to 3) indicate greater accuracy. The scores are summed to obtain an overall total that ranges from 0 to 9. Higher scores indicate the absence of asymmetry and greater precision in performance.
Catherine Bergego Scale (CBS) | The assessment is conducted within a week of admission to the ward.
  The Catherine Bergego Scale (CBS) is a clinical tool for measuring unilateral spatial neglect in patients with brain injuries, assessing how it impacts daily activities. The scale includes 10 activities (e.g., body orientation, mobility, personal care), each rated on a score from 0 to 3, where 0 indicates no neglect and 3 indicates severe neglect. The total score ranges from 0 to 30: higher scores indicate greater severity of neglect.
Visual neglect test | The assessment is conducted within a week of admission to the ward.
  Visual Field Testing: Assessing the ability to perceive visual stimuli in different quadrants can help identify neglect. Patients may be asked to report stimuli presented in specific visual fields, with significant omissions indicating neglect.
Mini Mental State Examination (MMSE) | During the assessment required for the neuropsychological evaluation of the patient, conducted as per standard clinical practice upon admission to the ward.
  (Range: 0-30; higher score=best performance).
Tactile neglect test | The assessment is conducted within a week of admission to the ward.
  Tactile Extinction Test: Patients are touched on both sides of the body simultaneously and must report where they feel the touch. If they can only report touch on one side when both sides are stimulated, it indicates tactile extinction and suggests neglect.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona - UOC di Neuroriabilitazione, Verona, verona, Italy